CLINICAL TRIAL: NCT06602869
Title: Cellular Markers During a Non-tuberculous Mycobacterial Respiratory Infection, Treated or Untreated, in Patients With Cystic Fibrosis
Brief Title: Cellular Markers in Treated or Untreated Non-tuberculous Mycobacterial Respiratory Infection in Patients With Cystic Fibrosis
Acronym: MUCEM
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Hôpital Cochin (Other); Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL24_0124
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Non-Tuberculous Mycobacterial Pneumonia
Keywords: Cystic Fibrosis; Interferon gamma release assay; Diagnostic Test
MeSH Terms: conditions — Cystic Fibrosis | interventions — myotrophin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case group MNT +: Cystic fibrosis patients with positive serology and positive culture
  Interventions: Other: Scheduled visit (V1)
- Control group MNT -: Cystic fibrosis patients with negative serology and negative culture
  Interventions: Other: Scheduled visit (V1)

INTERVENTIONS:
Other: Scheduled visit (V1) — During the scheduled visit (V1), as part of routine care, a blood draw will be performed. On this occasion, an additional 7 ml tube will be collected to perform serology and culture. This will help define the group (NTM+ Cases/NTM- Controls) and measure cellular biomarkers.

SUMMARY:
This study evaluates a diagnostic serological test for Non-Tuberculous Mycobacteria (NTM) infection in cystic fibrosis patients by measuring T cell response. It aims to highlight a dynamic response associated to the pathogen's presence. This multicenter case-control study involves two populations, providing a better understanding of the circulating T-IFNγ-MNT response in these patients.

DETAILED DESCRIPTION:
Background: Evidence shows that Non-tuberculous Mycobacterial (NTM) infections have increased and are 1,000 to 8,000 times more frequent in patients with cystic fibrosis compared to the general population. The diagnosis is based on clinical, radiological, and microbiological criteria. Unfortunately, the first two criteria lack specificity, and microbiological detection of NTM is limited due to frequent sputum contamination by other pathogens in cystic fibrosis patients. Given these factors and the high incidence of NTM infections in this population, alternative diagnostic methods are necessary.

Aim: This study aims to validate an innovative diagnostic test based on the IGRA (Interferon-Gamma Release Assay) method, which measures T lymphocyte response to Interferon gamma (IFNγ). The test will be conducted on a subset of patients selected from the CIMeNT cohort (ID-RCB: 2017-A00025-48). This cohort consists of cystic fibrosis patients whose NTM infection prevalence has been previously assessed.

Method: This research is a multicenter case-control study. It includes two groups: a case group of patients with positive serological and/or microbiological responses indicating NTM infection, and a control group of patients without such responses. The test measures the host's immune response by evaluating circulating T cell activity. Specifically, it measures IFNγ release when T cells are in contact with NTM antigens. This method provides more informative diagnostics of NTM infection dynamics compared to serology or microbiology, which have known technical limitations.

The study involves a single visit, which is part of the routine care for cystic fibrosis patients. During this visit, a routine blood draw will be performed and an additional 7 ml tube will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥18 years
* Patient previously included in the CIMeNT study
* Patient with a confirmed diagnosis of cystic fibrosis regardless of CFTR genotype
* Patient affiliated to the social security system
* Patient registered in the French Cystic Fibrosis Registry
* Adult patient capable of spontaneous expectoration or after induction

Exclusion Criteria:

* Lung transplant patients
* Person placed under judicial protection
* Pregnant and breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with cystic fibrosis included in the CIMeNT study (N°ID RCB : 2017-A00025-48)
Sampling Method: Non-Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-17 (Estimated)

PRIMARY OUTCOMES:
Determination of interferon-gamma release assay | day 1 (V1)
  Evaluation of T lymphocyte activation following mycobacterial antigen stimulation. The level of interferon gamma (IFN-γ) released is the measured marker of this activation, quantified in IU/ml. Sensitivity and specificity pairs will be calculated for each threshold value of the IFNγ rate in the T cell response test.
  A Receiver Operating Characteristic (ROC) curve will be plotted with its Area Under the Curve (AUC) and 95% confidence interval. For each threshold, sensitivity and specificity values will be computed, along with their 95% confidence intervals.
  The assessment aims to diagnose NTM in patients, as confirmed by serology and/or positive culture.

SECONDARY OUTCOMES:
Evaluation of T lymphocyte response | day 1 (V1)
  Measurement of IFN-γ release in response to T cell contact with NTM antigens, compared to clinical and radiological progression.

CONTACTS AND LOCATIONS:
Overall Officials: Raphael CHIRON, MD, Principal Investigator — Hôpital Arnaud de Villeneuve
Locations (1):
- CHU de Montpellier - Hôpital Arnaud de Villeneuve, Montpellier, France